CLINICAL TRIAL: NCT04077463
Title: An Open-label Phase 1/1b Study to Evaluate the Safety and Pharmacokinetics of JNJ-73841937 (Lazertinib), a Third Generation EGFR-TKI, as Monotherapy or in Combinations With JNJ-61186372, a Human Bispecific EGFR and cMet Antibody in Participants With Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of Lazertinib as Monotherapy or in Combination With Amivantamab in Participants With Advanced Non-small Cell Lung Cancer
Acronym: Chrysalis-2
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108656; 73841937NSC1001 (Other: Janssen Research & Development, LLC); 2020-000747-31 (EudraCT Number); 2023-506577-35-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib; amivantamab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Phase 1 (monotherapy dose escalation): Lazertinib (Experimental): Participants will receive Lazertinib monotherapy orally once daily (QD) in 21-day cycles until documented evidence of disease progression, unacceptable toxicity, noncompliance, or withdrawal of consent, or the investigator decides to discontinue treatment, whichever comes first. The subsequent doses of Lazertinib will be assigned by the Study Evaluation Team (SET) according to the dose escalation strategy by Bayesian logistic regression model (BLRM).
  Interventions: Drug: Lazertinib
- Phase 1b (combination): Lazertinib and Amivantamab (Experimental): Participants will receive Lazertinib and Amivantamab, after the safety of RP2D of Lazertinib is confirmed in the Phase 1, in 28-day cycles until documented evidence of disease progression, unacceptable toxicity, noncompliance, or withdrawal of consent, or the investigator decides to discontinue treatment, whichever comes first. This phase will start enrolling participants after the safety of Amivantamab is confirmed in Japanese participants in Study 61186372EDI1001 (NCT02609776).
  Interventions: Drug: Lazertinib; Drug: Amivantamab
- Phase 1b (combination): Lazertinib, Amivantamab and Platinum-doublet Chemotherapy (LACP) (Experimental): Participants will receive Lazertinib starting dose administered orally once daily (QD) in combination with Amivantamab, and doses of platinum-based chemotherapy (carboplatin and pemetrexed) per standard of care according to local guidance in a 21-day cycle for 4 cycles followed by maintenance with Lazertinib, Amivantamab and pemetrexed until disease progression or unacceptable toxicities.
  Interventions: Drug: Lazertinib; Drug: Amivantamab; Drug: Carboplatin; Drug: Pemetrexed
- Phase 1b (expansion) Cohort A: Lazertinib and Amivantamab (Experimental): This cohort A will further characterize the safety, tolerability, and preliminary antitumor activity of Lazertinib and Amivantamab based combinations within specific NSCLC population "who have progressed after osimertinib and subsequent platinum-based chemotherapy, and platinum-based chemotherapy regimen as the last line of therapy prior to study enrollment. Prior use of first or second generation EGFR TKI is allowed if administered prior to osimertinib. Participants will receive at the RP2CD of Lazertinib orally QD and Amivantamab, every 7 days for the first 28 days cycle and every 2 weeks thereafter.
  Interventions: Drug: Lazertinib; Drug: Amivantamab
- Phase 1b (expansion) Cohort B: Lazertinib and Amivantamab (Experimental): This Cohort B will further characterize the safety, tolerability and preliminary antitumor activity of Lazertinib and JNJ-61186372 combination in participants previously treated with advanced or metastatic NSCLC with documented primary EGFR Exon 20ins activating mutation. Participants will receive at the RP2CD of Lazertinib orally QD and Amivantamab, every 7 days for the first 28 days cycle and every 2 weeks thereafter.
  Interventions: Drug: Lazertinib; Drug: Amivantamab
- Phase 1b (expansion) Cohort C: Lazertinib and Amivantamab (Experimental): This Cohort C will further characterize the safety, tolerability and preliminary antitumor activity of Lazertinib and JNJ-61186372 combination in participants with uncommon EGFR mutations. Participants will receive at the RP2CD of Lazertinib orally QD and Amivantamab, every 7 days for the first 28 days cycle and every 2 weeks thereafter.
  Interventions: Drug: Lazertinib; Drug: Amivantamab
- Phase 1b (expansion) Cohort D: Lazertinib and Amivantamab (Experimental): Cohort D will seek to validate one or both potential biomarker strategies (next generation sequencing [NGS] and Immunohistochemical [IHC]), previously identified in Cohort E of Study 61186372EDI1001, in participants with osimertinib-relapsed, but chemotherapy-naive, EGFR Exon19del or L858R mutated NSCLC. Participants will receive at the RP2CD of Lazertinib orally QD and Amivantamab, every 7 days for the first 28 days cycle and every 2 weeks thereafter.
  Interventions: Drug: Lazertinib; Drug: Amivantamab
- Phase 1b (expansion) Cohort E: Lazertinib and Amivantamab (Experimental): Participants will receive at the RP2CD of Lazertinib orally QD and Amivantamab, every 7 days for the first 28 days cycle and every 2 weeks thereafter. Cohort E will seek to validate the immunohistochemical (IHC)-based biomarker strategy, by characterizing the activity of Amivantamab and Lazertinib combination in biomarker-positive participants with osimertinib-relapsed, but chemotherapy-naïve, EGFR Exon19del or L858R mutated NSCLC. In addition, Cohort E will seek to collect prospective data to confirm that prophylactic anticoagulation safely and effectively decreases the incidence of VTE events for patients treated with the combination of Amivantamab and Lazertinib, using Cohort F as reference.
  Interventions: Drug: Lazertinib; Drug: Amivantamab
- Phase 1b (expansion) Cohort F: Amivantamab Monotherapy (Experimental): Participants will receive Amivantamab monotherapy once weekly (QW) for 4 weeks, then every 2 weeks thereafter. Cohort F will seek to validate the IHC-based biomarker strategy, previously identified in Cohort D, by characterizing the activity of JNJ-61186372 monotherapy (Cohort F) in biomarker-positive participants with osimertinib-relapsed, but chemotherapy-naïve, EGFR Exon19del or L858R mutated NSCLC.
  Interventions: Drug: Amivantamab

INTERVENTIONS:
Drug: Lazertinib — Lazertinib will be administered orally.
  Other Names: JNJ-73841937
  Arms: Phase 1 (monotherapy dose escalation): Lazertinib; Phase 1b (combination): Lazertinib and Amivantamab; Phase 1b (combination): Lazertinib, Amivantamab and Platinum-doublet Chemotherapy (LACP); Phase 1b (expansion) Cohort A: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort B: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort C: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort D: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort E: Lazertinib and Amivantamab
Drug: Amivantamab — Amivantamab will be administered as an intravenous (IV) infusion.
  Other Names: JNJ-61186372
  Arms: Phase 1b (combination): Lazertinib and Amivantamab; Phase 1b (combination): Lazertinib, Amivantamab and Platinum-doublet Chemotherapy (LACP); Phase 1b (expansion) Cohort A: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort B: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort C: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort D: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort E: Lazertinib and Amivantamab; Phase 1b (expansion) Cohort F: Amivantamab Monotherapy
Drug: Carboplatin — Carboplatin will be administered as IV infusion.
  Arms: Phase 1b (combination): Lazertinib, Amivantamab and Platinum-doublet Chemotherapy (LACP)
Drug: Pemetrexed — Pemetrexed will be administered as IV infusion.
  Arms: Phase 1b (combination): Lazertinib, Amivantamab and Platinum-doublet Chemotherapy (LACP)

SUMMARY:
The purpose of this study is to confirm the tolerability of recommended Phase 2 dose (RP2D) of Lazertinib (Phase 1), to determine the tolerability and identify the recommended Phase 2 combination dose of Lazertinib when combined with Amivantamab (JNJ-61186372) (Phase 1b), to characterize the safety and tolerability of Lazertinib and Amivantamab combinations at the RP2CD in participants with advanced non-small cell lung cancer (NSCLC) with documented advanced or metastatic epidermal growth factor receptor (EGFR) mutation (Phase 1b expansion cohorts A, B, C, D and E), to estimate the antitumor activity of Lazertinib and Amivantamab combinations at the RP2CD in participants with advanced NSCLC with documented advanced or metastatic EGFR mutation (Phase 1b expansion cohorts A, B, C, and D), to validate the biomarker identified in Phase 1b expansion Cohort D as a predictor of antitumor activity of Lazertinib and Amivantamab combination (Cohort E) or Amivantamab monotherapy (Cohort F) in participants with osimertinib-relapsed, chemotherapy-naïve, EGFR Exon19del or L858R mutated NSCLC, to identify the recommended Phase 2 dose (RP2ChD) of Lazertinib when combined with Amivantamab and standard of care chemotherapy and to determine the tolerability of the Lazertinib, Amivantamab, and platinum-doublet chemotherapy (LACP) combination (Phase 1b LACP combination cohort) and to characterize the safety and tolerability of Lazertinib at the RP2ChD and Amivantamab and standard of care chemotherapy in participants with advanced or metastatic EGFR-mutated NSCLC (Phase 1b LACP combination cohort), to assess 2 potential biomarker strategies to identify participants at increased, or decreased, probability of tumor response with JNJ-61186372 and lazertinib combination in participants with EGFR Exon19del or L858R mutated NSCLC progressed on or after osimertinib (Phase 1b expansion Cohort D).

DETAILED DESCRIPTION:
Lung cancer is one of the most common types of cancer and is also the most common cause of death from cancer. NSCLC accounts for 85 percent (%) to 90% of lung cancers. Lazertinib is an oral, highly potent, mutant-selective, and irreversible EGFR-tyrosine kinase inhibitor (TKI) targeting both, the T790M mutation and activating EGFR mutations while sparing wild type EGFR. JNJ-61186372 (also referred to as amivantamab), is a low fucose, fully human immunoglobulin G1(IgG1)-based bispecific antibody. As a third generation EGFR-TKI targeting activating EGFR mutations, lazertinib has a distinct mechanism of action from JNJ-61186372, which targets the extracellular domains of both the EGFR and cMet proteins. The distinct mechanisms of action of lazertinib and JNJ-61186372 suggests potential to improve clinical outcomes through the combination of these two molecules. Phase 1 and 1b lazertinib + amivantamab, and Phase 1b LACP combination cohort are divided into 2 periods: screening and treatment period whereas Phase 1b expansion cohorts are divided into 3 periods: screening, treatment, and post-treatment follow up period. Safety assessment will include adverse events (AEs), serious adverse events (SAEs), physical examinations, Eastern Cooperative Oncology Group (ECOG) criteria for performance status, laboratory tests, vital signs, electrocardiograms, chest x-ray, baseline ophthalmologic examination (Phase 1b Expansion Cohorts), echocardiography or multigated acquisition, and concomitant medication usage. The overall duration of the study will be up to 5 years and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 and Phase 1b lazertinib+Amivantamab combination cohorts: Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) with previously epidermal growth factor receptor (EGFR) mutation (identified locally in a Clinical Laboratory Improvement Amendments [CLIA]-certified laboratory [or equivalent]) that is metastatic or unresectable, and have progressed after standard of care front-line therapy, and exhausted available options with targeted therapy. A participant who has refused all other currently available therapeutic options is allowed to enroll
* For the Phase 1b Lazertinib, Amivantamab and Platinum-doublet Chemotherapy (LACP) combination cohort: histologically or cytologically confirmed advanced or metastatic EGFR-mutated NSCLC who have progressed on or after an EGFR-TKI as the most recent line of treatment with a maximum of 3 prior lines of therapy in the metastatic setting allowed
* For all expansion cohorts, the EGFR mutation must have been previously histologically or cytologically characterized, as performed by a CLIA-certified (US sites) or an accredited (outside of US) local laboratory, with a copy of the mutation analysis being submitted during screening (Phase 1b expansion Cohort B, C, D, E, and F)

  1. Expansion Cohort A: Participant must have advanced or metastatic EGFR-mutated non-small cell lung cancer (NSCLC) that has progressed on prior treatment with osimertinib in the first or second line, followed by progression on a platinum-based chemotherapy regimen as the last line of therapy prior to study enrollment. Prior use of first or second generation EGFR tyrosine kinase inhibitor (TKI) is allowed if administered prior to osimertinib
  2. Expansion Cohort B: Participant must have previously treated, advanced or metastatic NSCLC with documented primary EGFR Exon 20ins activating mutation. Participants should have been treated with standard of care, platinum-based chemotherapy regimens, but may have treated with approved EGFR TKI, investigational EGFR, or immunotherapy agents if refusing front line platinum-based chemotherapy standard of care. Up to 3 lines of prior systemic anti-cancer treatment are allowed
  3. Expansion Cohort C: Participant must have advanced or metastatic NSCLC characterized by an uncommon activating mutation Additional uncommon EGFR mutations/alterations, beyond those listed above, may be considered for enrollment after agreement with the medical monitor. Participants may be treatment naïve or have been treated with one prior line of therapy which must be a first or second generation TKI (that is gefitinib, erlotinib, afatinib) in the most recent line of therapy. Prior chemotherapy is allowed if administered prior to EGFR TKI therapy, or as the only systemic anti-cancer therapy prior to study enrollment. Up to 2 lines of prior systemic anti-cancer treatment are allowed
  4. Expansion Cohort D, E, and F: Participant must have advanced or metastatic EGFR-mutated NSCLC (EGFR Exon19 deletion or L858R) that has progressed on prior treatment with osimertinib in the first or second line (after first- or second-generation EGFR TKI), as the immediate prior line of therapy. Only previous treatment in the metastatic setting with a first, second, or third generation EGFR TKI is allowed. In addition, participants considered for Cohorts E and F must be eligible for, and agree to comply with, the use of prophylactic anticoagulation with a direct oral anticoagulant or a low molecular weight heparin during the first 4 months (from Day 1 through Day 120) according to national comprehensive cancer network (NCCN) or local guidelines, if assigned to the combination Cohort E
* Evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Participants must meet the study protocol defined laboratory criteria without having a history of red blood cell transfusion, platelet transfusion, or granulocyte-colony stimulating factor support within 7 days prior to the date of the test
* A woman of childbearing potential: Must have a negative serum beta human chorionic gonadotropin at screening; Must agree not to breast-feed during the study and for 6 months after the last dose of study intervention. (Enrollment is not allowed even if a woman who is breast-feeding stops breast-feeding); Must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study intervention

Exclusion Criteria:

* Participant has an uncontrolled illness, including but not limited to uncontrolled diabetes, ongoing or active infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week prior to study treatment] or diagnosed or suspected viral infection); active bleeding diathesis; Impaired oxygenation requiring continuous oxygen supplementation; Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of study treatment; or psychiatric illness or any other circumstances (including social circumstances) that would limit compliance with study requirements. Any ophthalmologic condition that is either clinically unstable or requires treatment
* Prior treatment with anti programmed cell death-1 (PD-1) or anti programmed cell death-ligand 1 (PD-L1) antibody within 6 weeks of planned first dose of study intervention
* Untreated brain or other central nervous system (CNS) metastases whether symptomatic or asymptomatic. Participants who have completed definitive therapy, are not on steroids, and have a stable clinical status for at least 2 weeks prior to study treatment may be eligible for Phase 1b expansion cohorts. If brain metastases are diagnosed on Screening imaging, the participant may be enrolled, or rescreened for eligibility, after definitive treatment if above criteria are met
* Any Toxicities from prior anticancer therapy must have resolved to common terminology criteria for adverse events (CTCAE) version 5.0 Grade 1 or baseline level (except for alopecia [any grade], Grade <=2 peripheral neuropathy, and Grade <=2 hypothyroidism stable on hormone replacement therapy)
* Allergies, hypersensitivity, or intolerance to Lazertinib or JNJ-61186372 or their excipients. For the LACP combination cohort: participant has a contraindication for the use of carboplatin or pemetrexed (refer to local prescribing information for each agent). Participant has a history of hypersensitivity to, or cannot take, vitamin B12 or folic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2028-03-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicity (DLT) (Phase 1) | Until the end of first cycle (21 days for Phase 1)
  DLTs are defined as certain non-hematologic and hematologic toxicities of Grade 3 or higher.
Percentage of Participants with Dose-Limiting Toxicity (DLT) (Phase 1b) | Until the end of first cycle (28 days for Phase 1b)
  DLTs are defined as certain non-hematologic and hematologic toxicities of Grade 3 or higher.
Overall Response Rate (ORR) (Phase 1b Expansion Cohorts A-D) | Up to 2.5 years
  ORR is defined as the percentage of participants who achieve either a complete (CR) or partial response (PR) as determined by the investigator using RECIST 1.1 criteria.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability (Phase 1b Expansion Cohorts A-E) | Up to 2.5 years
  Adverse events (AEs) defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Criteria Version 5.0 in participants treated at the RP2CD regimen of Lazertinib and Amivantamab combination therapy. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Percentage of Participants with DLT (Phase 1b combination Lazertinib, Amivantamab, Platinum-doublet chemotherapy [LACP]) | Until the end of first cycle (21 days for Phase 1b combination LACP)
  DLTs are defined as certain non-hematologic and hematologic toxicities of Grade 3 or higher.
Number of Participants with AEs as a Measure of Safety and Tolerability (Phase 1b combination LACP) | Up to 2.5 years
  AEs defined by the NCI-CTCAE criteria version 5.0 in participants treated with LACP combination regimen. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Overall Response Rate (ORR) per RECIST version 1.1 (v1.1) with NGS Analysis of Circulating Tumor ctDNA, IHC Analysis of EGFR and MET Expression (Phase 1b Expansion Cohort D) | Up to 2.5 years
  ORR is defined as the percentage of participants who achieve either a complete (CR) or partial response (PR) as determined by the investigator using RECIST 1.1 criteria with Next Generation Sequencing (NGS) Analysis of Circulating Tumor Deoxyribonucleic Acid (ctDNA), Immunohistochemical (IHC) Analysis of Tumor Epidermal Growth Factor Receptor (EGFR) and MET Expression (Phase 1b Expansion Cohort D).
ORR Among Participants with MET3+ Staining on Greater Than or Equal to (>=)25 Percent (%) of Tumor Cells (Phase 1b Expansion Cohorts E and F) | Up to 2.5 years
  ORR among participants with MET3+ staining on >=25 % of tumor cells will be reported. ORR is defined as the percentage of participants who achieve either a CR or PR as determined by the investigator using RECIST 1.1 criteria.
Duration of Response (DOR) Among Participants with MET3+ Staining on >=25% of Tumor Cells (Phase 1b Expansion Cohorts E and F) | Up to 2.5 years
  DOR among participants with MET3+ staining on >=25 % of tumor cells will be reported. DOR will be calculated as time from initial response of CR or PR to progressive disease (PD) or death due to any cause, whichever comes first, only for participants who achieve CR or PR as determined by the investigator using RECIST 1.1 criteria.
Clinical Benefit Rate (CBR) Among Participants with MET3+ Staining on >=25% of Tumor Cells (Phase 1b Expansion Cohorts E and F) | Up to 2.5 years
  CBR among participants with MET3+ staining on >=25% of tumor cells will be reported. CBR is defined as the percentage of participants achieving complete or partial response, or durable stable disease (duration of at least 11 weeks) as determined by the investigator using RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability (Phase 1 and Phase 1b) | Up to 2.5 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Plasma Concentration of Lazertinib (Phase 1 and Phase 1b) | Up to End of Treatment [EOT]) (30 days after last dose) (up to 2.5 years)
  Plasma samples will be analyzed to determine concentrations of Lazertinib.
Serum Concentration of Amivantamab (Phase 1b) | Up to EOT (30 days after last dose) (up to 2.5 years)
  Serum samples will be analyzed to determine concentrations of Amivantamab.
Number of Participants with Anti-drug Antibodies Against Amivantamab (Phase 1b) | Up to EOT (30 days after last dose) (up to 2.5 years)
  Number of participants with anti-drug antibodies against Amivantamab will be reported.
Progression free survival (PFS) (Phase 1b Expansion) | Up to 2.5 years
  PFS is defined as the time from first infusion of study intervention to PD or death due to any cause.
Time to Treatment Failure (TTF) (Phase 1b Expansion) | Up to 2.5 years
  TTF is defined as the time from the first administration of the study intervention to discontinuation of treatment for any reason, including disease progression, treatment toxicity, death, and will be utilized to capture clinical benefit for patients continuing treatment beyond as determined by the investigator using RECIST 1.1 criteria.
Overall Survival (OS) (Phase 1b Expansion) | Up to 2.5 years
  OS is defined as the time from first infusion of study intervention to death due to any cause as determined by the investigator using RECIST 1.1 criteria.
Duration of Response (DOR) (Phase 1b expansion) | Up to 2.5 years
  DOR will be calculated as time from initial response of CR or PR to progressive disease (PD) or death due to any cause, whichever comes first, only for participants who achieve CR or PR as determined by the investigator using RECIST 1.1 criteria.
Clinical Benefit Rate (CBR) (Phase 1b expansion) | Up to 2.5 years
  CBR is defined as the percentage of participants achieving complete or partial response, or durable stable disease (duration of at least 11 weeks) as determined by the investigator using RECIST 1.1 criteria.
Number of Participants with Venous Thromboembolic (VTE) Events by Severity | Up to 2.5 years
  Number of participants with VTE events including pulmonary embolism and deep vein thrombosis by severity defined by the NCI-CTCAE Criteria Version 5.0 will be reported.
Number of Participants with Adverse Events (AEs) (Phase 1b Expansion Cohort F) | Up to 2.5 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
ORR (Phase 1b expansion Cohorts E and F) | Up to 2.5 years
  ORR is defined as the percentage of participants who achieve either a CR or PR as determined by the investigator using RECIST 1.1 criteria.
DOR (Phase 1b Expansion Cohorts E and F) | Up to 2.5 years
  DOR will be calculated as time from initial response of CR or PR to PD or death due to any cause, whichever comes first, only for participants who achieve CR or PR as determined by the investigator using RECIST 1.1 criteria.
CBR (Phase 1b expansion Cohorts E and F) | Up to 2.5 years
  CBR is defined as the percentage of participants achieving complete or partial response, or durable stable disease (duration of at least 11 weeks) as determined by the investigator using RECIST 1.1 criteria.
Intracranial Progression free survival (PFS) (Phase 1b Expansion E and F) | Up to 2.5 years
  Intracranial PFS is defined as the time from first infusion of study intervention until the date of objective intracranial disease progression or death, whichever comes first, based on Investigator assessment using RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (78):
- United States (18):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Irvine, Orange, California
  - UCSF Helen Diller Comprehensive, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Cedars Sinai Medical Center, West Hollywood, California
  - H. Lee Moffitt Cancer & Research Institute, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Langone Health at NYC University, NYU School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania Division of Hematology Oncology Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington, Seattle, Washington
- China (14):
  - Beijing Cancer Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Hunan Cancer hospital, Changsha
  - West China School of Medicine/West China Hospital, Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Central Hospital of Jinan, Jinan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - Shanghai Chest Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- France (7):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Institut Curie, Paris
  - CHU De Poitiers, Poitiers
  - HIA Begin, Saint-Mandé
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Evangelische Lungenklinik Berlin, Berlin
  - Uniklinik Köln, Cologne
  - Kliniiken der Stadt Köln gGmbH, Krankenhaus Köln-Mehrheim, Cologne
  - Universitaetsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - Asklepios Klinik Gauting GmbH - Asklepios Fachkliniken Munchen-Gauting, Gauting
  - Städtisches Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle
  - Lungenklinik Hemer, Hemer
  - Pius-Hospital Oldenburg, Oldenburg
  - Robert-Bosch-Krankenhaus - Klinik Schillerhoehe, Stuttgart
- Italy (5):
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Istituto Europeo di Oncologia, Milan
  - San Gerardo Hospital, Monza
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Ospedale S. Maria Delle Croci, Ravenna
- Japan (7):
  - National Cancer Center Hospital, Chūōku
  - Kansai Medical University Hospital, Hirakata
  - National Cancer Center Hospital East, Kashiwa
  - Kobe City Medical Center General Hospital, Kobe
  - Aichi Cancer Center Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Shizuoka Cancer Center, Shizuoka
- Oncologic Hospital, Puerto Rico Medical Center, Rio Piedras, Puerto Rico
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp. Virgen Del Rocio, Seville
- Taiwan (4):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency